CLINICAL TRIAL: NCT05548413
Title: Improving Medication Adherence Using Family-focused and Literacy-sensitive Strategies in Patients With Heart Failure
Brief Title: Improving Medication Adherence Using Family-focused and Literacy-sensitive Strategies
Acronym: FamLit_HF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jia-Rong Wu (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor-Investigator, Jia-Rong Wu, Associate Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 80203; 1R01NR020478-01 (NIH)
Record Dates: First submitted 2022-09-16; First posted 2022-09-21 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Medication Adherence; Heart Failure
Keywords: care partner; family; health literacy; teach back
MeSH Terms: conditions — Medication Adherence; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patients - Attention Only (Active Comparator): Patients with a confirmed diagnosis of heart failure.
  Interventions: Behavioral: Attention Control
- Care Partners - Attention Only (Active Comparator): Care partners of patients with a confirmed diagnosis of heart failure.
  Interventions: Behavioral: Attention Control
- Patients - FamLit (Experimental): Patients with a confirmed diagnosis of heart failure.
  Interventions: Behavioral: FamLit
- Care Partners - FamLit (Experimental): Care partners of patients with a confirmed diagnosis of heart failure.
  Interventions: Behavioral: FamLit

INTERVENTIONS:
Behavioral: FamLit — The FamLit (Family-focused and Literacy-sensitive strategy) is an interactive, multi-component intervention supported by the FamLit intervention Guide, including both spoken and printed materials written at a 4th-grade reading level for HF patients and their primary CPs.Three constructs guide the intervention, based on the Theory of Planned Behavior (TPB): 1) develop patient and CP positive attitudes through HF instruction and teach-back; 2) form positive subjective norms through coaching to improve patient and CP communication, support, and teamwork; and 3) increase perceived behavioral control through coaching and role-playing to empower patients and CPs to overcome individual barriers to adherence. This intervention also includes use of the SimpleMed+ electronic pillbox.
  Arms: Care Partners - FamLit; Patients - FamLit
Behavioral: Attention Control — Participants in this group will talk with an interventionist to discuss general health. This intervention also includes use of the SimpleMed+ electronic pillbox.
  Arms: Care Partners - Attention Only; Patients - Attention Only

SUMMARY:
People with heart failure who do not take their medications as prescribed are at high risk of complications leading to hospitalization, death and poor quality of life. In the proposed intervention, nurses will use easy-to-understand language to coach patients and their care partners to help them work together and build skills to overcome their individual barriers to adherence in order to 1) improve and sustain patient medication adherence; 2) reduce hospitalization; 3) improve quality of life. If effective, this intervention will support long-term medication adherence, thus reducing hospitalizations related to heart failure and quality of life.

DETAILED DESCRIPTION:
Medication adherence is thought by many providers and researchers to be the most important self-care behavior, yet it is also the most problematic. Poor medication adherence can cause poor quality of life (QoL), hospitalization, and death. In the United States, approximately 125,000 deaths per year are due to poor medication adherence and up to 50% of heart failure (HF) patients are re-hospitalized within 6 months of a previous HF exacerbation and one of the most common causes is poor medication adherence. Lifelong and usually complex medication regimens are needed for patients with HF, yet 40-60% of HF patients have suboptimal medication adherence. Health literacy plays a significant role in suboptimal medication adherence. Support by a care partner (CP; usually a family member) can improve adherence and reduce hospitalizations. Although some interventions have improved HF patients' adherence, improvements were small, and effects were not sustained. To enhance and sustain intervention effects, an approach that is literacy-sensitive and incorporates social support will be used. Using easy-to-understand language for patients and CPs, investigators will test an interactive, behavioral, family-focused and literacy-sensitive (FamLit) intervention delivered by nurses, incorporating evidence-based, multi-components (e.g., teach-back, coaching, role-playing, goal setting) to engage both patients and CPs in improving and sustaining medication adherence and health outcomes. A randomized controlled trial will be conducted to evaluate the efficacy of FamLit intervention on medication adherence, hospitalization, death, and QoL. 164 dyads of patients and their primary CPs (patients-CPs) will be randomly assigned to either the FamLit intervention or an attention-control group. Both groups will have an in-person session (delivered on the day of a clinic appointment for regular follow-up) one month after baseline and phone boosters every other week for up to 3 months. FamLit group sessions will focus on improving medication adherence, and control group sessions will focus on general health issues. Aims are to: 1) test the efficacy of the FamLit intervention compared to an attention control group on outcomes (i.e., primary: medication adherence, and secondary: a) HF hospitalization or all-cause death, b) QoL over 12 months.

ELIGIBILITY:
Inclusion Criteria - Patient Participants:

* confirmed diagnosis of heart failure (HF), either systolic or diastolic HF
* ave suboptimal medication adherence
* have a care partner (CP) (either spouse, daughter/son, partner, other relative, friend) who is identified by the patient as the person most involved in HF care
* willingness to have a CP be involved in their medication taking
* have undergone evaluation of HF and prescribed stable doses of HF medications for at least 3 months
* live in a setting where the patient is responsible for their ow medication administration
* willing to use the SimpleMed+ (i.e., an electronic pillbox to measure objective medication adherence)
* availability by phone

Exclusion Criteria - Patient Participants:

* cognitive impairment as indicated by having difficulties to understand and give informed consent
* a recent hospitalization within 3 months of study enrollment
* co-existing end-stage renal disease or terminal illness such as advanced malignancy, or any other condition with less than 1-year life expectancy
* psychotic illness
* current alcohol dependence or other substance abuse
* inability to speak English or other communication barrier
* currently or have received any similar self-care intervention recently in the past year

Inclusion Criteria - Care Partners:

* unpaid family member, friend, partner, or other relation who is involved in the patients' care at least 3 times a week, designated by the patient
* willing to receive interventions with the patient together
* 18 years of age or older

Exclusion Criteria - Care Partners:

* cognitive impairment as indicated by having difficulties to understand and give informed consent
* coexisting terminal illness
* non-English speaking or any other communication barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2023-01-04 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Medication adherence | 12 months
  Percentage of prescribed doses taken (PDT%) as determined by the electronic SimpleMed+ pillbox. SimpleMed+ will record the date and time that the lid of each compartment is opened and closed. Those data will be used to calculate objective medication adherence: percent prescribed doses taken (PDT%) = (# of doses taken during monitoring period)/(# of prescribed doses during monitoring period) x 100.PDT% ranges from 0-100%.
Self-reported medication adherence. | 12 months
  Adherence will be surveyed the Basel Assessment of Adherence Scale (BAAS), a copyrighted, self-reported scale. The BAAS includes 5 yes-no items and one visual analogue scale (VAS). If participants indicate they have missed a dose (a "yes" response) to any of 5 dichotomous items and <80% on the VAS, they are classified as suboptimally medication adherent.

SECONDARY OUTCOMES:
Patient hospitalization | 12 months
  Percentage of patients hospitalized. HF hospitalizations will be determined by a combination of medical record review and monthly phone interviews with patients and/or care partners to collect data for all encounters.
Quality of life - Minnesota Living with Heart Failure | 12 months
  The 21-item Minnesota Living with Heart Failure (MLHF) questionnaire measures the patient's perceptions of the influence of HF on physical and emotional aspects of life. The items are scored on a Likert scale from 0 (No) to 5 (Very much). The scores of the 21 items will be summed with higher scores of the MLHF indicating worse quality of life.
Positive Affect | 12 months
  Generic quality of life will be assessed using the NeuroQoL Positive Affect and Well-Being short form, which has 9 items and each item is rated on a 5-point Likert scale from 1 (never) to 5 (always); higher scores indicate better quality of life.

OTHER OUTCOMES:
Caregiver Burden | 12 months
  The Zarit Caregiver Burden Interview (ZBI) measures caregiver burden. The ZBI has 12 items and each item is rated on a 5-point Likert scale from 0 (never) to 4 (always); higher scores indicate higher caregiver burden.
Numeracy health literacy | 12 months
  The Newest Vital Sign (NVS) will be used to assess numeracy. Participants will be given a nutritional label and be asked 6 questions about its content. Participants will get one point for each question they are correct. Participants will be scored on the number of questions they get correct, higher scores indicate better numeracy health literacy.
Health Literacy | 12 months
  The 36-item Short Test of Functional Health Literacy in Adults (S-TOFHLA),which has 36-items. Participants will be scored on the number of items they got correct (one point for each correct item), higher scores indicate better health literacy. Patients and CPs will be categorized as low (0-22) or high (23-36) health literacy.
Medication Adherence Scale | 12 months
  The psychometrically sound Medication Adherence Scale (MAS) with 3 subscales to measure constructs of the Theory of Planned Behavior. The Attitude subscale has 7 items on a Likert scale from 0 (strongly disagree) to 10 (strongly agree), higher scores indicate better attitudes. The Subjective Norm subscale has 4 items on a Likert scale from 1 (strongly disagree) to 5 (strongly agree), higher scores indicate more positive subjective norm. The Perceived Behavioral Control subscale has 12 items on a Likert scale from 0 (never being a cause) to 10 (very important cause), higher scores indicate more barriers.
Communication | 12 months
  Communication will be measured using the 6-item Family Assessment Device (FAD) Communication subscale. Each survey item is scored on a Likert scale from 1 (strongly disagree) to 4 (strongly agree). The FAD is scored by adding the responses (1-4) of the 6 items and dividing by 6. Higher scores indicate worse levels of family functioning on communication.
Social Support | 12 months
  We will assess social support using the 8-item, modified Medical Outcome Study Social Support Scale (mMOS-SS). Each survey item is scored on a Likert scale from 1 (none of the time) to 5 (all of the time). The total sum of the items is then used to calculate a mMOS-SS score with values between 0 and 100, with higher scores indicating better social support.

CONTACTS AND LOCATIONS:
Overall Officials: Jia-Rong Wu, Principal Investigator — University of Kentucky
Locations (1):
- Jia-Rong Wu, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No